CLINICAL TRIAL: NCT07090421
Title: Varying Doses of Evening Caffeine Ingestion Have Different Effects on Rowing Ergometer Performance, Sleep Quality and Wakefulness Scores
Brief Title: Caffeine Dose: Performance and Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulaç Can YILDIRIM (Other)
Responsible Party: Sponsor-Investigator, Ulaç Can YILDIRIM, Assoc. Prof., Sinop University
Organization: Sinop University (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2021/80
Record Dates: First submitted 2025-07-04; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Healthy Volunteers; Caffeine; Sleep Quality
Keywords: Caffeine; Dose-response; Rowing performance; Sleep quality; Wakefulness
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Caffeine; Powders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Participants ingested an inert cellulose capsule containing no active substance approximately 60 minutes prior to performing a 2000-meter rowing ergometer time trial. This condition served as the control to compare the effects of caffeine ingestion at varying doses.
  Interventions: Dietary Supplement: Cellulose Powder
- Low Dose Caffeine (Experimental): Participants ingested a caffeine capsule at a dosage of 3 mg per kg of body mass approximately 60 minutes before the 2000-meter rowing ergometer trial. This condition was included to evaluate the ergogenic and sleep-related effects of a low evening caffeine dose.
  Interventions: Dietary Supplement: Caffeine 3 mg/kg Oral Powder
- Moderate Dose Caffeine (Experimental): Participants ingested a caffeine capsule at a dosage of 6 mg per kg of body mass approximately 60 minutes before performing the 2000-meter rowing ergometer test. This condition represented a commonly used moderate dose to examine its impact on performance and sleep parameters.
  Interventions: Dietary Supplement: Caffeine 6 mg/kg Oral Powder
- High Dose Caffeine (Experimental): Participants ingested a caffeine capsule at a dosage of 9 mg per kg of body mass approximately 60 minutes prior to the rowing trial. This high-dose condition was used to assess the maximum ergogenic potential of caffeine and its possible detrimental effects on sleep quality and next-day recovery.
  Interventions: Dietary Supplement: Caffeine 9 mg/kg Oral Powder

INTERVENTIONS:
Dietary Supplement: Cellulose Powder — Participants consumed an inert cellulose powder dissolved in water, containing no active caffeine. The placebo was ingested orally 60 minutes prior to the rowing performance test. This condition served as the control and was administered once per session in a randomized, double-blind, crossover design.
  Arms: Placebo
Dietary Supplement: Caffeine 3 mg/kg Oral Powder — Participants consumed caffeine in powder form at a dose of 3 milligrams per kilogram of body weight. The powder was dissolved in water and ingested orally approximately 60 minutes before the start of the 2000-meter rowing ergometer performance test. The intervention was administered once per session in a randomized, double-blind, crossover design.
  Arms: Low Dose Caffeine
Dietary Supplement: Caffeine 6 mg/kg Oral Powder — Participants ingested caffeine in powder form, dissolved in water, at a dose of 6 milligrams per kilogram of body mass. The solution was consumed orally 60 minutes prior to the 2000-meter rowing performance test. This intervention was administered once per session as part of a randomized, double-blind, crossover design.
  Arms: Moderate Dose Caffeine
Dietary Supplement: Caffeine 9 mg/kg Oral Powder — A powdered caffeine dose of 9 milligrams per kilogram was dissolved in water and consumed orally by participants 60 minutes before a 2000-meter rowing ergometer trial. The intervention was administered once per session under a randomized, double-blind, crossover design.
  Arms: High Dose Caffeine

SUMMARY:
The goal of this clinical trial is to learn how different doses of caffeine taken in the evening affect rowing performance, sleep quality, and daytime alertness in trained male university rowers. The main questions it aims to answer are:

Does a low, moderate, or high caffeine dose improve rowing performance? How do these doses affect sleep and recovery after evening exercise? Participants completed four rowing tests after consuming either a placebo, low (3 mg/kg), moderate (6 mg/kg), or high (9 mg/kg) dose of caffeine. Researchers measured rowing time, power, heart rate, sleep quality, and daytime sleepiness.

The study found that moderate and high caffeine doses improved rowing performance the most. However, these same doses made it harder for participants to sleep well and feel alert the next day. Headaches and stomach issues were also more common with the high dose. The low dose gave smaller performance gains but caused fewer side effects.

This study shows that evening caffeine can boost performance but may hurt recovery and sleep. Athletes and coaches should weigh these trade-offs when using caffeine for late-day training or competition.

DETAILED DESCRIPTION:
This double-blind, randomized crossover study examined the dose-dependent effects of evening caffeine ingestion on rowing performance, sleep quality, and daytime alertness in trained male university rowers. The rationale stems from increasing use of caffeine as a performance-enhancing supplement in evening training or competition settings, despite its known adverse effects on sleep and recovery. Thirteen participants completed four experimental trials (placebo, 3 mg/kg, 6 mg/kg, 9 mg/kg caffeine), each separated by a washout period, during which they performed a 2000-meter rowing time trial and were assessed for sleep quality and daytime sleepiness using validated scales. The study also recorded physiological responses and adverse events across conditions. By evaluating multiple doses, the design allowed for assessment of both efficacy and tolerability thresholds, supporting dose-optimization strategies. This study aims to inform practical guidelines for athletes and coaches balancing acute ergogenic benefits with potential recovery trade-offs when caffeine is used late in the day.

ELIGIBILITY:
Inclusion Criteria:

* Male university-level rowers
* Aged approximately 22 ± 2.2 years
* Minimum of 2 years of rowing training experience
* Free of any medical condition that impairs exercise participation
* Regular caffeine consumers (habitual daily intake recorded)
* Voluntarily signed informed consent form
* Available to attend all scheduled laboratory sessions

Exclusion Criteria:

* Any medical condition that could interfere with study participation or protocol adherence
* Use of prescription medications during the study period
* Known allergy to mannitol or other artificial sweeteners
* Diagnosed sleep disorders (e.g., insomnia, sleep apnea)
* Physician's advice to limit or avoid caffeine intake

Ages: 20 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2022-07-24 (Actual); Primary Completion 2022-08-24 (Actual); Study Completion 2022-08-24 (Actual)

PRIMARY OUTCOMES:
Change in 2000-meter Rowing Ergometer Completion Time (seconds) Following Varying Doses of Evening Caffeine Ingestion | Approximately 60 minutes post-ingestion on each test day, during evening sessions (between 6:00 PM and 9:00 PM)
  The time in seconds required to complete a 2000-meter rowing ergometer trial was recorded under four separate conditions: placebo, and caffeine doses of 3 mg/kg, 6 mg/kg, and 9 mg/kg. Each participant completed one trial per condition in a randomized, double-blind, crossover design. Performance was measured using a Concept2 rowing ergometer with integrated time-tracking software. Trials were conducted in the evening (between 6:00 PM and 9:00 PM), approximately 60 minutes after ingestion of the assigned supplement. A lower time indicates better performance.
Subjective Sleep Quality Score (5-point Likert Scale) | Morning following each test day (approximately 10-12 hours post-dose)
  Participants rated their perceived sleep quality the morning after each trial using a 5-point Likert scale (1 = very poor, 5 = very good). Scores reflect subjective assessment of sleep quality following evening caffeine ingestion.
Mean Power Output (Watts) During 2000-meter Rowing Ergometer Trial | Approximately 60 minutes post-ingestion on each test day, during evening sessions (between 6:00 PM and 9:00 PM)
  Average power output (in watts) generated by participants during each 2000-meter rowing trial. Power was recorded via Concept2 ergometer's internal performance monitor, calculated over the full distance. A higher value indicates better performance.
Daytime Sleepiness Score (Epworth Sleepiness Scale) | Morning following each test day (approximately 10-12 hours post-dose)
  Daytime sleepiness was assessed using the Epworth Sleepiness Scale (ESS), a validated questionnaire consisting of 8 items, each scored from 0 to 3. Total scores range from 0 (no sleepiness) to 24 (severe sleepiness). Higher scores indicate more sleepiness.

CONTACTS AND LOCATIONS:
Overall Officials: Ulas C. Yildirim, pHd, Principal Investigator — Sinop University
Locations (1):
- Sinop University Facility, Sinop, Centarl, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) underlying the results reported in the publication, including performance outcomes, sleep-related metrics, and adverse event reports, will be made available upon reasonable request to qualified researchers. Data will be de-identified to protect participant confidentiality. The data will become accessible after publication of the main results and will be available for up to five years. A data dictionary will also be provided to facilitate proper interpretation.
Supporting Information: Study Protocol, SAP
Time Frame: Individual participant data (IPD) will be available beginning 6 months after publication of the study results and will be accessible for up to 5 years.
Access Criteria: Qualified researchers who provide a methodologically sound proposal will be granted access to the deidentified individual participant data. Proposals should be submitted to [your email address or institutional contact]. Access will be granted for research purposes only and in accordance with data use agreements.

REFERENCES:
- [Background] Ali A, O'Donnell JM, Starck C, Rutherfurd-Markwick KJ. The Effect of Caffeine Ingestion during Evening Exercise on Subsequent Sleep Quality in Females. Int J Sports Med. 2015 Jun;36(6):433-9. doi: 10.1055/s-0034-1398580. Epub 2015 Feb 20. PMID 25700100
- [Background] Anderson ME, Bruce CR, Fraser SF, Stepto NK, Klein R, Hopkins WG, Hawley JA. Improved 2000-meter rowing performance in competitive oarswomen after caffeine ingestion. Int J Sport Nutr Exerc Metab. 2000 Dec;10(4):464-75. doi: 10.1123/ijsnem.10.4.464. PMID 11099373
- [Background] Bonnar D, Bartel K, Kakoschke N, Lang C. Sleep Interventions Designed to Improve Athletic Performance and Recovery: A Systematic Review of Current Approaches. Sports Med. 2018 Mar;48(3):683-703. doi: 10.1007/s40279-017-0832-x. PMID 29352373
- [Background] Chen B, Ding L, Qin Q, Lei TH, Girard O, Cao Y. Effect of caffeine ingestion on time trial performance in cyclists: a systematic review and meta-analysis. J Int Soc Sports Nutr. 2024 Dec;21(1):2363789. doi: 10.1080/15502783.2024.2363789. Epub 2024 Jun 5. PMID 38836626
- [Background] de Souza JG, Del Coso J, Fonseca FS, Silva BVC, de Souza DB, da Silva Gianoni RL, Filip-Stachnik A, Serrao JC, Claudino JG. Risk or benefit? Side effects of caffeine supplementation in sport: a systematic review. Eur J Nutr. 2022 Dec;61(8):3823-3834. doi: 10.1007/s00394-022-02874-3. Epub 2022 Apr 5. PMID 35380245
- [Background] Drapeau C, Hamel-Hebert I, Robillard R, Selmaoui B, Filipini D, Carrier J. Challenging sleep in aging: the effects of 200 mg of caffeine during the evening in young and middle-aged moderate caffeine consumers. J Sleep Res. 2006 Jun;15(2):133-41. doi: 10.1111/j.1365-2869.2006.00518.x. PMID 16704567

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-24): https://cdn.clinicaltrials.gov/large-docs/21/NCT07090421/Prot_SAP_000.pdf